CLINICAL TRIAL: NCT03405961
Title: A Single-site Self-controlled Comparative Study of Conventional Versus Digital Peer Assessment Rating (PAR) Using the Carestream (CS) 3600 Intraoral Scanner in Orthodontic Patients
Brief Title: A Comparison of Conventional Versus Digital PAR (Peer Assessment Rating) Scores Using an Intraoral Scanner
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Kingston Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 230630
Record Dates: First submitted 2017-12-18; First posted 2018-01-23 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Malocclusion
Keywords: PAR scoring; Digital study models
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Manual PAR score: Patient will receive upper and lower impressions, which will be cast to produce plaster models. A calibrated individual will PAR score the casts in the traditional manner (regular care pathway)
- Direct digital PAR score: Patient will receive upper and lower intra-oral scans which will be PAR scored directly by the computer
  Interventions: Device: Carestream 3600 intra oral scan
- Indirect digital PAR score: Patient will receive upper and lower impressions which will be cast to produce plater models (regular care pathway). The casts will be scanned with Carestream 3600 intra oral scanner and scored digitally by the computer.
  Interventions: Device: Carestream 3600 intra oral scan

INTERVENTIONS:
Device: Carestream 3600 intra oral scan — Carestream 3600 is CE marked intra oral scanner manufactured by Carestream Dental. It is already licensed for use in dentistry to produce digital study models. The scanner is 220 x 38 x 58 mm large and operates using video capture technology. It emits no radiation.
  Carestream 3600 is connected to a computer via a USB port and a computer software (CS Model +) converts the scan into digital study models using trigonometric calculations. The software is then used to take measurements on the digital models and calculate PAR scores
  Groups: Direct digital PAR score; Indirect digital PAR score

SUMMARY:
In dentistry, Peer Assessment Rating (PAR) is an objective way of quantifying how maligned a patient's teeth are by scoring orthodontic study models. It can also be used to assess treatment outcome by comparing pre- and post-treatment scores. Traditionally, PAR scoring is performed manually on plaster casts by a trained and calibrated individual. The plaster casts consume considerable amounts of storage space and the process of manual scoring can be time consuming and expensive. The recent decades have seen a rise in popularity of intra oral scanners in dentistry to produce digital study models. These obviate the need for physical storage space and a software can be used to calculate PAR scores more conveniently and at a faster speed. A review of the current literature showed that the CS 3600 intra oral scanner by Carestream Dental demonstrated acceptable accuracy for clinical use.

In this study, patients will receive the usual impressions and their moulds will be PAR scored manually (usual care pathway). In addition, they will also receive intra oral scans with Carestream 3600 and the digital models will be scored by a computer. Manual and digital scores will be compared and analysed for any significant discrepancies.

DETAILED DESCRIPTION:
CS 3600 intra oral scanner is already licenced for the use in dentistry and is routinely used by some dental practitioners to substitute conventional impressions and plaster models in restorative, implant and orthodontic diagnosis and treatment planning. The scanner is 220 x 38 x 58 mm in size and operates with video capture technology. It emits no radiation.

Peer Assessment Rating (PAR) is an objective way of quantifying how severe a malocclusion is by scoring orthodontic study models. It can also be used to assess treatment outcome. All National Health Service (NHS) orthodontic providers in the United Kingdom are contractually bound to submit PAR score changes for at least 20 of their treated cases plus 10% of the remainder of their case load every year. Traditionally, PAR scoring is performed manually on plaster casts by a trained and calibrated individual. The plaster casts must be retained as part of the patient's medical records and hence consume considerable amounts of storage space. The process of manual scoring is also time intensive. Digital models obviate the need for physical storage space and a software can be used to calculate PAR scores more conveniently and at a faster speed. A review of the current literature showed that the CS 3600 intra oral scanner by Carestream Dental demonstrated acceptable accuracy for clinical use. The purpose of this study is to assess the accuracy of PAR scores obtained from digital models with those obtained manually from conventional models for the same patient at one given point in time.

Aims: Against this background, the aim of this study is to compare digital PAR scoring using the CS 3600 intraoral scanner with conventional PAR scoring.

Objectives: The objectives are to investigate whether PAR scoring on models acquired through direct and indirect digitisation produces any significant errors when compared with conventional PAR scoring on plaster models. The study will also seek to measure the chairside time taken to produce upper and lower full arch scans and bite registration with CS 3600 versus the time taken to produce equivalent alginate impressions and wax bite. Furthermore, the time taken for digital scoring will be measured and compared with the conventional method. Finally, patient preference with regard to intraoral scans versus impressions will be investigated.

Method: The sample size was confirmed using a power calculation. The sample will consist of 66 orthodontic patients at Kingston Hospital, excluding any patients with fixed appliances or bonded components. All patients will receive conventional impressions as well as intraoral scans, serving as their own controls. Plaster casts poured from the impressions will also be scanned to produce indirect digital models. PAR scoring will then be performed by one investigator on all three models (plaster casts, direct and indirect digital models) for comparison. A second investigator will record the time taken to perform scans and impressions as well as the time taken to complete digital and conventional scoring. Immediately after the clinical procedure patients will be given a questionnaire evaluating their preference.

Data analysis: Data from the PAR scorings and questionnaires will be recorded and analysed using SPSS following consultation with a bio-statistician. The data will then be graphically represented in the form of tables and charts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing orthodontic treatment at Kingston Hospital
2. Patients who have completed their orthodontic treatment and are attending for retainer reviews at Kingston Hospital
3. age 11-50

Exclusion Criteria:

1. patients with fixed or bonded appliances
2. age <11 or >50
3. Inability to gain informed consent due to communication barriers

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: orthodontic patients at Kingston Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Peer Assessment Rating (PAR) score | 6 months
  PAR score is an objective and standardised way of quantifying how much the position of teeth deviate from an ideal. Sub-scores are given in 5 categories assessing the position of teeth to adjacent teeth in same jaw as well as the opposing jaw. The sub scores are weighted according to their importance as described by Richmond et al. (1992) and then added to give a total score. Total scores may range from 2 to approximately 50. The higher the score, the greater the deviation from ideal.

SECONDARY OUTCOMES:
The length of time (in minutes) taken to obtain conventional impressions | 6 months
  The time taken to take conventional impressions (from insertion into the mouth until removal from the mouth) will be measured using a stop watch. The time taken to create digital impressions (from activating the scanner until completion of the scan, including any areas that need to be re-scanned) will also be measured using a stop watch.
The length of time (in minutes) taken to obtain digital scans | 6 months
  The time taken to take conventional impressions (from insertion into the mouth until removal from the mouth) will be measured using a stop watch. The time taken to create digital impressions (from activating the scanner until completion of the scan, including any areas that need to be re-scanned) will also be measured using a stop watch.
The cost involved in creating digital scans | 6 months
  In order to calculate the cost of conventional models, the sum of the following will be calculated: cost of impression material (the amount of impression material used will be recorded), cost of impression tray, cost of tray adhesive, disinfection cost, laboratory and transport cost.
  In order to calculate the cost of digital impressions, the sum of the following will be calculated: cost of scanner and software, cost of disposable scanner tip covers
The cost involved in creating conventional models | 6 months
  In order to calculate the cost of conventional models, the sum of the following will be calculated: cost of impression material (the amount of impression material used will be recorded), cost of impression tray, cost of tray adhesive, disinfection cost, laboratory and transport cost.
  In order to calculate the cost of digital impressions, the sum of the following will be calculated: cost of scanner and software, cost of disposable scanner tip covers
Do patients prefer conventional impressions or intraoral scans? | 6 months
  This will be assessed by means of a questionnaire consisting of 3 validated questions. The questions are designed to establish which of the two procedures the patient found 1. more comfortable, 2. quicker and 3. which they would prefer to undergo again.

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Cobourne, BDS MOrth, Principal Investigator — King's College London
Locations (1):
- Kingston Hospital, Kingston upon Thames, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only pseudonymised data will be shared. No patient identifiable material will be shared with other researchers.

REFERENCES:
- [Derived] Luqmani S, Jones A, Andiappan M, Cobourne MT. A comparison of conventional vs automated digital Peer Assessment Rating scoring using the Carestream 3600 scanner and CS Model+ software system: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2020 Feb;157(2):148-155.e1. doi: 10.1016/j.ajodo.2019.10.011. PMID 32005465